CLINICAL TRIAL: NCT02678988
Title: A Study to Evaluate the Bioequivalence of Tocilizumab Following Subcutaneous Administration Via an Autoinjector (AI 1000-G2) Versus a Pre-Filled Syringe in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: WA30003
Record Dates: First submitted 2016-02-08; First posted 2016-02-10 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — tocilizumab

ARMS (6):
- A1: Tocilizumab AI followed by PFS-NSD in abdomen (Experimental): Participants will receive two single doses of 162 milligrams (mg) tocilizumab SC, first dose via AI on Day 1 (Period 1) followed by a washout period of 6 weeks, thereafter second dose via PFS-NSD on Day 43 (Period 2), in abdomen.
  Interventions: Device: AI-1000 G2; Device: PFS-NSD; Drug: Tocilizumab
- A2: Tocilizumab AI followed by PFS-NSD in thigh (Experimental): Participants will receive two single doses of 162 mg tocilizumab SC, first dose via AI on Day 1 (Period 1) followed by a washout period of 6 weeks, thereafter second dose via PFS-NSD on Day 43 (Period 2) in thigh.
  Interventions: Device: AI-1000 G2; Device: PFS-NSD; Drug: Tocilizumab
- A3: Tocilizumab AI followed by PFS-NSD in upper arm (Experimental): Participants will receive two single doses of 162 mg tocilizumab SC, first dose via AI on Day 1 (Period 1) followed by a washout period of 6 weeks, thereafter second dose via PFS-NSD on Day 43 (Period 2), in upper arm.
  Interventions: Device: AI-1000 G2; Device: PFS-NSD; Drug: Tocilizumab
- B1: Tocilizumab PFS-NSD followed by AI in abdomen (Experimental): Participants will receive two single doses of 162 mg tocilizumab SC, first dose via PFS-NSD on Day 1 (Period 1) followed by a washout period of 6 weeks, thereafter second dose via AI on Day 43 (Period 2), in abdomen.
  Interventions: Device: AI-1000 G2; Device: PFS-NSD; Drug: Tocilizumab
- B2: Tocilizumab PFS-NSD followed by AI in thigh (Experimental): Participants will receive two single doses of 162 mg tocilizumab SC, first dose via PFS-NSD on Day 1 (Period 1) followed by a washout period of 6 weeks, thereafter second dose via AI on Day 43 (Period 2), in thigh.
  Interventions: Device: AI-1000 G2; Device: PFS-NSD; Drug: Tocilizumab
- B3: Tocilizumab PFS-NSD followed by AI in upper arm (Experimental): Participants will receive two single doses of 162 mg tocilizumab SC, first dose via PFS-NSD on Day 1 (Period 1) followed by a washout period of 6 weeks, thereafter second dose via AI on Day 43 (Period 2), in thigh.
  Interventions: Device: AI-1000 G2; Device: PFS-NSD; Drug: Tocilizumab

INTERVENTIONS:
Device: AI-1000 G2 — The device will contain TCZ (180 milligrams per milliliter [mg/mL]) SC formulation single dose of 0.9 mL that corresponds to 162 mg TCZ administered via PFS and assembled in the AI (AI-1000 G2).
Device: PFS-NSD — The device will contain TCZ (180 mg/mL) SC formulation single dose of 0.9 mL that corresponds to 162 mg TCZ administered via PFS-NSD.
Drug: Tocilizumab — Participants will receive two single doses of 162 mg tocilizumab SC on Day 1 (Period 1) and Day 43 (Period 2), with a washout period of 6 weeks between the periods.
  Other Names: RO4877533; Actemra/RoActemra

SUMMARY:
The study consists of an eligibility screening period, two study periods involving single doses of tocilizumab (TCZ) according to an open-label, randomized, two-period crossover design with an interval of 6 weeks between periods, and a 6 week follow-up period. Healthy participants will receive a single subcutaneous (SC) injection of TCZ via a pre-filled syringe-needle safety device (PFS-NSD) and a single injection via an autoinjector (AI). The total duration of the study is up to 16 weeks from screening to follow-up. After screening, eligible participants will be randomly assigned to one of the two possible treatment sequences (Sequence 1: AI-1000 G2 followed by PFS-NSD or Sequence 2: PFS-NSD followed by AI-1000 G2) and assigned to one of three injection sites (1: abdomen, 2: thigh, or 3: upper arm). All participant groups will receive a total of two TCZ administrations each.

ELIGIBILITY:
Inclusion Criteria:

* Male participants and their partners of child-bearing potential must be willing to use two effective contraceptive methods
* Female participants must be either postmenopausal or surgically sterile
* Intact normal skin in the area for intended injection
* Body weight less than (<) 150 kilograms (kg)
* Have no contraindications from the following: a detailed medical and surgical history, a complete physical examination, including vital signs, 12-lead electro cardio gram (ECG), hematology, blood chemistry, serology, and urinalysis

Exclusion Criteria:

* Participants with any known active current or history of recurrent Infectious disease
* Positive result on hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus-1 (HIV-1) and HIV-2 at screening
* A history of clinically significant gastrointestinal, renal, hepatic, cardiovascular, or allergic disease
* Evidence of malignant disease, or malignancies diagnosed within the previous 5 years
* Use of or being dependent within the last 12 months on any substances of abuse, including a relevant past history of alcohol abuse
* Participants with a history of, or currently active primary or secondary immunodeficiency
* Participants who smoke more than 10 cigarettes per day or equivalent in tobacco
* Clinically relevant deviation from normal in the physical examination, including vital signs
* Clinically relevant ECG abnormalities on screening
* Evidence of atrial fibrillation, atrial flutter, right or left bundle branch block, Wolf-Parkinson-White syndrome, or cardiac pacemaker or any other significant cardiac abnormalities
* Known allergy to TCZ or any other ingredient in the subcutaneous (SC) formulation
* History of severe allergic or anaphylactic reactions to human, humanized, or murine monoclonal antibodies
* Known coagulopathy
* Clinically significant abnormalities in laboratory test results
* Immunization with a live or attenuated vaccine is prohibited within 4 weeks prior to study drug administration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2016-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Maximum observed serum concentration (Cmax) of TCZ | Pre-dose and 8 hours post-dose on Day 1, and pre-dose on Days 2, 3, 4, 5, 6, 8, 10, 13, 16, 19, 22, 29, 36, pre-dose and 8 hours post-dose on Day 43, and pre-dose on Days 44, 45, 46, 47, 48, 50, 52, 55, 58, 61, 64, 71, 78 and 85
Area under the serum concentration-time curve from time zero to last quantifiable concentration (AUClast) of TCZ | Pre-dose and 8 hours post-dose on Day 1, and pre-dose on Days 2, 3, 4, 5, 6, 8, 10, 13, 16, 19, 22, 29, 36, pre-dose and 8 hours post-dose on Day 43, and pre-dose on Days 44, 45, 46, 47, 48, 50, 52, 55, 58, 61, 64, 71, 78 and 85

SECONDARY OUTCOMES:
Area under the serum concentration-time curve from time zero to extrapolated infinite time [AUC (0-inf)] of TCZ | Pre-dose and 8 hours post-dose on Day 1, and pre-dose on Days 2, 3, 4, 5, 6, 8, 10, 13, 16, 19, 22, 29, 36, pre-dose and 8 hours post-dose on Day 43, and pre-dose on Days 44, 45, 46, 47, 48, 50, 52, 55, 58, 61, 64, 71, 78 and 85
Time to reach maximum observed serum concentration (Tmax) of TCZ | Pre-dose and 8 hours post-dose on Day 1, and pre-dose on Days 2, 3, 4, 5, 6, 8, 10, 13, 16, 19, 22, 29, 36, pre-dose and 8 hours post-dose on Day 43, and pre-dose on Days 44, 45, 46, 47, 48, 50, 52, 55, 58, 61, 64, 71, 78 and 85
Apparent elimination rate constant (Kel) of TCZ | Pre-dose and 8 hours post-dose on Day 1, and pre-dose on Days 2, 3, 4, 5, 6, 8, 10, 13, 16, 19, 22, 29, 36, pre-dose and 8 hours post-dose on Day 43, and pre-dose on Days 44, 45, 46, 47, 48, 50, 52, 55, 58, 61, 64, 71, 78 and 85
Number of participants with adverse events | Baseline up to 8 weeks after the last dose of study drug (approximately 7 months)
Number of participants with anti-drug antibody (ADA) response | Pre-dose on Days 1 and 43, and Day 85

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- United States (3):
  - Lenexa, Kansas
  - Marlton, New Jersey
  - Salt Lake City, Utah

REFERENCES:
- [Derived] Fettner S, Mela C, Wildenhahn F, Tavanti M, Wells C, Douglass W, Mallalieu NL. Evidence of bioequivalence and positive patient user handling of a tocilizumab autoinjector. Expert Opin Drug Deliv. 2019 May;16(5):551-561. doi: 10.1080/17425247.2019.1604678. Epub 2019 May 2. PMID 31043095